CLINICAL TRIAL: NCT02091531
Title: A Phase 2 Study of the Dual mTOR Inhibitor MLN0128 in Patients With Metastatic Castration-Resistant Prostate Cancer (CRPC)
Brief Title: Dual mTOR Inhibitor MLN0128 in Advanced Castration-Resistant Prostate Cancer (CRPC) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-143
Record Dates: First submitted 2014-03-14; First posted 2014-03-19 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2018-10

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: mTOR Inhibitor MLN0128; PSA; 13-143
MeSH Terms: interventions — sapanisertib

ARMS (1):
- MLN0128 (Experimental): Patients will be treated with the established phase II dose of MLN0128 (4mg po daily continuously; 1 cycle=4 weeks) to assess mechanisms of sensitivity and resistance in men with CRPC who have received either enzalutamide and/or abiraterone.
  Interventions: Drug: MLN0128

INTERVENTIONS:
Drug: MLN0128

SUMMARY:
This is a phase II study which will test the study drug MLN0128 in patients with castration resistant prostate cancer who have received chemotherapy in the past. Phase II clinical trials test how well an investigational drug works in treating a specific cancer. "Investigational" means that the drug is still being studied and that research doctors are trying to find out more about it. MLN0128 is not approved by the FDA.

The purpose of this study is to see what effects (good and bad) the study drug MLN0128 has on the patient and the cancer. MLN0128 is a drug that belongs to a class of drugs called "mTOR kinase inhibitors". A protein, called "mTOR" inside the cells in the body, plays a role in controlling how cells grow. In some cancer cells, mTOR may be over-active. This over-activity may cause some cancer cells to grow out of control. Research has shown that mTOR inhibitors can block this overactivity and may help stop or slow down the growth of some types of cancer cells.

ELIGIBILITY:
To be included in this study, patients should have histologically confirmed castration resistant metastatic prostate cancer with evidence of disease progression. Patients must have been in a castrate state either by orchiectomy or by GnRH analogues. In detail, they should meet all of the following criteria

Inclusion Criteria:

* Histologically confirmed prostate cancer with progressive metastatic disease based on any of the following: i) a rise in PSA, ii) transaxial imaging, or iii) radionuclide bone scan.

  1. PSA - a minimum of 3 consecutive rising levels, with an interval of ≥

     1 week between each determination. The last determination must have a minimal value of ≥ 2 ng/mL and be determined within two weeks prior to enrollment.
  2. Measurable Disease - patients showing new or progressive soft tissue masses on CT or MRI scans as defined by the PCWG2 criteria21
  3. Radionuclide bone scan - at least two new metastatic lesions.
* Detectable metastases by bone scan, CT-scan or MRI.
* Ongoing androgen depletion therapy with a Gonadotropin Releasing Hormone (GnRH) analogue or inhibitor, or orchiectomy (i.e., surgical or medical castration).

For patients who have not had an orchiectomy, there must be a plan to maintain effective GnRH-analogue therapy for the duration of the trial.

* Castrate levels of serum testosterone < 50 ng/dL determined within 4 weeks prior to starting treatment.
* Patients who are receiving an anti-androgen as part of their first-line hormonal therapy must have shown progression of disease off the anti-androgen prior to enrollment.
* At least 4 weeks must have elapsed from the use of androgen receptor antagonists (i.e., flutamide, nilutamide, bicalutamide, enzalutamide ); 5-α reductase inhibitors (i.e., finasteride, aminoglutethimide); abiraterone acetate; estrogens; nitrosoureas, mitomycin C, isotype therapy, ketoconazole, chemotherapy and other anti-cancer pharmacologic therapy prior to beginning protocol therapy.
* At least 8 weeks must have elapsed from the use of Strontium-89, Radium-223, Samarium-153, or immunotherapy (e.g., Provenge) prior to beginning protocol therapy.
* At least 4 weeks must have elapsed from the use of any investigational agent prior to beginning protocol therapy.

  a. Note: Prior treatment with PI3K/mTOR pathway inhibitors prohibited.
* At least 4 weeks must have elapsed from major surgery.
* Toxicities related to prior therapy must either have returned to ≤ Grade 1, baseline or deemed irreversible.
* Patients with treated, non-progressive epidural disease are eligible.
* KPS performance status 70-100% (50-60% is allowed only if due to bone pain)
* At least 18 years of age, with a life expectancy at least 3 months.
* Patient must be willing to comply with study procedures.
* Physical and laboratory test findings

  1. Adequate hepatic function with serum bilirubin ≤ 1.5 times the upper institutional limits of normal (ULN), ALT and AST ≤ 2.5 x ULN. Patients with a history of Gilbert's syndrome may be enrolled if the total bilirubin is < 3 mg/dL with a predominance of indirect bilirubin
  2. Adequate renal function with serum creatinine ≤ 1.5 x ULN.
  3. Adequate hematologic function with absolute neutrophil counts ≥ 1,500 cell/mm3 and platelets ≥ 100,000 cells/mm3 and hemoglobin value ≥ 9 g/dL (Note: patients whose anemia has been corrected to a hemoglobin value ≥ 9 g/dL with blood transfusions are allowed).
  4. Electrolytes (including potassium, sodium, and serum calcium corrected for albumin or ionized calcium) must be within normal limits.
* Left ventricular ejection fraction (LVEF) no more than 5 absolute percentage points below the institutional standard of normal as measured by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA) within 4 weeks prior to first study drug administration (ie, if the institutional normal is 50%, subject's LVEF may be as low as 45% to be eligible for the study)

Exclusion Criteria:

Patients that meet any of the criteria listed below will not be eligible for study entry:

* History of, or current known metastases in the brain or untreated spinal cord compression;
* History of another malignancy within the previous 2 years except for the following:

  1. Adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer,
  2. Adequately treated Stage I or II cancer currently in complete remission, or any other cancer that has been in complete remission for at least 2 years;
* Prior treatment with PI3K/mTOR pathway inhibitors;

Diabetes mellitus on active treatment, or subjects with either of the following:

1. Fasting blood glucose (FBG) ≥ 126 mg/dL (7.0 mmol/L), or
2. HbA1c ≥ 6.5%;

   * Use of herbal products that may decrease PSA levels (i.e., saw palmetto) or systemic corticosteroid greater than the equivalent of 10 mg of prednisone per day during the 4 weeks prior to screening or plans to initiate treatment with the above during the entire duration of the study;
   * Any history of unstable angina, myocardial infarction, New York Heart Association (NYHA) Class III or IV heart failure, and/or pulmonary hypertension;
   * Significant active cardiovascular disease including:

a. Uncontrolled high blood pressure (ie, systolic blood pressure > 180 mmHg, diastolic blood pressure > 95 mmHg) b. Grade 3 or higher valvular disease c. Grade 3 or higher atrial fibrillation d. Grade 3 or higher bradycardia e. Endocarditis f. Pulmonary embolism g. Recent cerebrovascular accident within 6 months prior to enrollment

* A requirement for positive inotropic support (excluding digoxin) or serious uncontrolled cardiac arrhythmia (including atrial flutter/fibrillation) within 1 year prior to screening
* A pacemaker or implantable cardiac defibrillator
* Known history of infection with human immunodeficiency virus (HIV), based on medical history (screening labs to rule out HIV infection are not required);
* Any other condition that, in the opinion of the Investigator, would impair the patient's ability to comply with study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-03; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Rathkopf, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- MLN0128: Patients will be treated with the established phase II dose of MLN0128 (4mg po daily continuously; 1 cycle=4 weeks) to assess mechanisms of sensitivity and resistance in men with CRPC who have received either enzalutamide and/or abiraterone.
  MLN0128
Period: Overall Study
Arm/Group | MLN0128
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MLN0128
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 67 [52 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Median Time on Treatment
Description: from the start of treatment, as defined by the Prostate Cancer Working Group 2 (PCWG2) guidelines.
Time Frame: Up to 8 months
Measure: Median (Full Range); unit: weeks
Arm/Group | MLN0128
Number analyzed (Participants) | 9
weeks | 11 [3 to 30]

2. Secondary Outcome: Median PSA Rise at End of Treatment as Compared to Baseline
Description: Summary tables and waterfall plots describing change in PSA relative to baseline will be reported at end of treatment
Time Frame: Duration of Treatment, up to 30 weeks
Measure: Median (Full Range); unit: percentage PSA increase from basline
Arm/Group | MLN0128
Number analyzed (Participants) | 9
percentage PSA increase from basline | 159 [12 to 620]

3. Secondary Outcome: Best Response
Description: We propose to study both FDG and optional FDHT PET imaging at baseline, 4 weeks after treatment initiation and at the time of progression (end-of-treatment), and to correlate the changes with treatment response. Response and progression will be evaluated in this study using a combination of the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee and modified for prostate cancer and the guidelines for prostate cancer endpoints developed by the Prostate Cancer Clinical Trials Working Group (PCWG2).21
Time Frame: Duration of Treatment, up to 30 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MLN0128
Number analyzed (Participants) | 9
Participants
  Stable Disease | 8
  Progression of Disease | 1

ADVERSE EVENTS:
Time Frame: Up to 8 months
Arm/Group | MLN0128
All-Cause Mortality (participants affected / at risk) | 9/9
Serious Adverse Events (participants affected / at risk) | 6/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLN0128 (N=9)
Allergic reaction (Immune system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Buttock Pain (Musculoskeletal and connective tissue disorders) | 1
Delirium (Product Issues) | 1
Dizziness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Edema limbs (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Platelet count decreased (Investigations) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MLN0128 (N=9)
Urinary frequency (Renal and urinary disorders) | 8
Fatigue (General disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 7
Mucositis (Gastrointestinal disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 9
Constipation (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 7
Pain (General disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Edema (General disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 2
Delirium (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT02091531/Prot_SAP_000.pdf